CLINICAL TRIAL: NCT00403026
Title: Off-Label,Intravitreal Use of Bevacizumab for Retinal Disorders
Brief Title: Intravitreal Bevacizumab for Retinal Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Narayana Nethralaya (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN-002/2006
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Last update posted 2006-11-23 (Estimated); Status verified 2006-11

CONDITIONS: Wet AMD; Macular Oedema; Proliferative Diabetic Retinopathy
Keywords: Bevacizumab (Avastin); Intravitreal injection; VEGF; CRVO; BRVO; PDR; CNVM
MeSH Terms: conditions — Macular Edema | interventions — Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab ( Avastin)

SUMMARY:
Bevacizumab is an anti-VEGF agent used in approved for use in metastatic colorectal carcinoma (FDA Approved). This study analyzes the safety and efficacy of off-label Intravitreal Injection of bevacizumab (Avastin) for CNVM, Macular oedema due to diabetic retinopathy, vascular occlusion and other retinal disorders.

DETAILED DESCRIPTION:
Purpose: To study the efficacy and safety of invitreal injection of bevacizumab (avastin) in all the following conditions.

* Age related macular degeneration with Juxtafoveal and Subfoveal CNVM: Recurrent CNVM following PDT and TTT with IVTA. Patient who could not afford PDT, Macugen or Lucentis which is FDA approved.
* Myopic CNVM, Idiopathic CNVM, Inflammatory CNVM and other conditions associated with CNVM.
* Refractory macular oedema due to vein occlusion, Pseudophakia, Clinically significant macular oedema (CSME) etc. that affects vision and does not respond adequately to usual treatment methods.
* Proliferative diabetic retinopathy, non-resolving vitreous haemorrhage with PDR
* Informed consent were taken from all the patients, based on the guidelines of OMIC (Ophthalmic mutual insurance company)Avastin: Risk management recommendations and consent form.

American Academy of ophthalmology-Risk management recommendations for off-label , Intravitreal use of Avastin.

Included indications, exclusion criteria, possible complications and the off-label status of the drug.

Best corrected visual acuity, Fundus Photography, anterior segment examination, Optical coherence tomography and in selected patients Electrophysiology, VEP and Fundus fluorescein angiography was done according to surgeons discretion.

All the patients were examined on day 1, 1st week and subsequently depending on the surgeons discretion and tests were performed during follow ups.

During follow up best-corrected visual acuity, anterior and posterior segment examination. Fundus photography, Intraocular pressure and OCT was repeated and in selected patients FFA, ERG,and VEP was done, physicians follow up was done.

Preparation of the Drug:

Bevacizumab Avastin (Avastin) comes in a sterile vial (100 mg in 4 ml) preservative free and ensure safety the vial injection was within a day.

Injections were given with 30 gauge needle, tuberculin syringes single use. 0.05ml containing 1.25 mg drug was given intravitreally under all aseptic precautions under topical anaesthesia,suggested by Flynn , Harry w.and scott, Ingrid u. -Evolving guidelines for intravitreous injections.

Following the injection topical antibiotics was given for 1 week.

Design: Prospective interventional non randomised case series.

Informed consent process

Informed consent was taken in English and the patients were explained in their local language by the treating surgeon.

The Food and Drug Administration approved Avastin for the treatment of metastatic Colorectal cancer. It is the first humanized Anti-VEGF antibody, which prevents angiogenesis. Since the drug is FDA approved the off-label drug is used for Intravitreal usage. For other purposes if patients are well-informed about the product, base, its use on firm scientific method and sound medical evidence, and maintain records of its use and effects. Ophthalmologists are using Avastin "off-label" to treat AMD and similar conditions since research indicates that VEGF is one of the causes for the growth of the abnormal vessels that cause these conditions. All the patients were informed about the "off-label" status, which is not FDA approved. Similar to kenalog, which is FDA approved but the off-label drug is used as Intravitreal injection to treat eye conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age related macular degeneration with Juxtafoveal and Subfoveal CNVM: Recurrent CNVM following PDT and TTT with IVTA. Patient who could not afford PDT, Macugen or Lucentis which is FDA approved.
* Myopic CNVM, Idiopathic CNVM, Inflammatory CNVM and other conditions associated with CNVM.
* Refractory macular oedema due to vein occlusion, Pseudophakia, Clinically significant macular oedema (CSME) etc. that affects vision and does not respond adequately to usual treatment methods.
* Proliferative diabetic retinopathy, non-resolving vitreous haemorrhage with PDR.

Exclusion Criteria:

* Patients with poor compliance
* Patients with uncontrolled diabetes and hypertension or any other medical condition that increase the risk of complications like recent history of Stroke or myocardial infraction (< one year). (Physician clearance was obtained for all patients).
* Patients who had undergone major surgery 28 days before, were excluded from the study and it was also suspended prior to elective surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2006-08; Study Completion 2006-11

PRIMARY OUTCOMES:
Vision change
Anatomical changes (Regression of NVE, CNVM, reduction in macular thickness)
Electrophysiological changes (ERG, VEP)

SECONDARY OUTCOMES:
Ocular side effects (infection, RD, IOP rise, cataract)

CONTACTS AND LOCATIONS:
Overall Officials: sivakami pai, MS, Principal Investigator — Narayana Nethralaya, Bangalroe, India
Locations (1):
- Sivakami Pai, Bangalore, India